CLINICAL TRIAL: NCT05057390
Title: Evaluating the Tolerance, Compliance, Acceptability and Safety of a New Human Milk Fortifier (NHMF) in Preterm Infants: a Case Study Series
Brief Title: HMF Preterm Case Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NHMF2020
Record Dates: First submitted 2021-09-06; First posted 2021-09-27 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Preterm Infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New Human Milk Fortifier (Experimental): From the Baseline (start of intervention) each patient will receive the case study product for at least 4 weeks (28 days), with at least 1-week administration in the community.
  Interventions: Dietary Supplement: New Human Milk Fortifier (NHMF)

INTERVENTIONS:
Dietary Supplement: New Human Milk Fortifier (NHMF) — The case study product will be added to human milk during the hospitalization and will continue after discharge for at least 1 week (7 days), to obtain community data. NHMF prescription will be specified on an individual basis by the investigating Dietitian responsible for the infant's nutritional management. The intervention period will end when the infant does not require NHMF (according to local neonatal guidelines and/or clinical indication).
  The case study product will be labelled specifically for the case study and will be available in a powder format.
  Full preparation, storage and safety instructions will be given to the parent/caregiver by the investigating Dietitian before commencing the case study product to ensure its correct and safe use.

SUMMARY:
Nutritional requirements in preterm infants can be elevated, as a result of complex clinical circumstances including infections, immaturity of the gastrointestinal tract and invasive treatments, such as surgery which can place a greater metabolic demand on the body. Furthermore, these circumstances can impact an infant's ability to meet nutritional requirements and achieve optimum growth through normal feeding alone. Most preterm infants may need specialist care by the neonatal team during hospital admission and post-discharge, which includes enteral nutritional support.

Human Milk Fortifier (HMF) have become a component of the routine clinical care of preterm infants on neonatal units. There is published evidence to support this practice as being safe and effective. A multitude of trials have demonstrated improvements in weight, length and head circumference following interventions using HMF, compared to non-supplemented cohorts, and benefits have been observed at long term follow up.

Whilst HMF is used routinely in neonatal units, there is little clinical evidence for using them beyond discharge in the community, although this is widely accepted in practice. Nutricia have developed a new HMF (NHMF) that can be provided for use in the community.

This series of case-studies will evaluate the tolerance, compliance, acceptability and safety of the NHMF, in 15 preterm infants. Each case study will last at least 28 days, including at least 7 days in the community setting. The case studies will be conducted across multiple specialist neonatal centres in the UK, to meet the UK ACBS requirements.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants fed own mother's milk (or donor human milk) requiring HMF (as decided by the investigator)
* Born before 37 weeks completed gestational age and >1 dropped centile since birth requiring HMF (as decided by the investigator)
* Tolerating adequate volume of enteral nutrition
* Expected to require HMF after discharge (minimum 4.0g NHMF per day at discharge)
* Written or electronic informed consent from parent/caregiver

Exclusion Criteria:

* Anticipated short term use of HMF leading to discontinuation of HMF after hospital discharge
* Presence of any relevant proven or suspected chromosomal anomaly or genetic syndrome, any gastrointestinal malformation/compromise, including Necrotising enterocolitis (NEC) (defined as Bell's stage two or higher), metabolic disorder, or congenital central nervous system malformation that may impact tolerance of enteral feeding
* Failure to establish enteral nutrition and requiring full parenteral nutrition
* Participation in other studies within 1 month prior to the entry of this study
* Known allergy to any of the study product ingredients, including cow's milk, fish and egg
* Concern or issues around the breast milk supply from mother of preterm infant at enrolment
* Investigator concerns around willingness/ability of the parent/caregiver to comply with protocol requirements and/or handle and store NHMF appropriately

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Gastro-intestinal tolerance | Baseline (Start of intervention) - End of case study (4 weeks administration)
  Gastro-intestinal (GI) tolerance will be recorded by the investigating Dietitian at the above-mentioned time-points. GI tolerance will be recorded using a standardised questionnaire, to be completed by the investigating Dietitian with the parent/caregiver, as appropriate. Parents/caregivers will be asked to recall the infant's symptoms in the past 24 hours to the investigating Dietitian, and as an average over the case study period, at each assessment point.

SECONDARY OUTCOMES:
Compliance | Baseline (Start of intervention) - End of case study (4 weeks administration)
  Compliance with the recommended intake during the case study period will be assessed by the investigating Dietitian at the above-mentioned time-points. The investigating Dietitian will ask parents/caregivers how much case study product was taken by the infant in the past 24 hours and on average over the case study period at each assessment. This will be compared to the amount prescribed by the Dietitian for the infant to consume daily which will be recorded at the start of the case study and any changes during the case study will be noted.
Anthropometrics | Baseline (Start of intervention) - End of case study (4 weeks administration)
  Growth of infants will be determined according to standardised procedures at the above-mentioned time-points. Body weight (grams) will be measured using a weighing scale. Length and head circumference will be measured to the nearest 0.1cm with a length board and non-stretchable tape measure respectively. Growth outputs will be plotted using UK Neonatal and Infant Close Monitoring Growth Charts to track changes over time. Actual growth will be compared to growth expectations set by the investigating Dietitian at the start of the case study (baseline)
Safety (adverse events) | Baseline (Start of intervention) - End of case study (4 weeks administration)
  All adverse events will be recorded throughout the case study

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Stratton, Study Chair — Nutricia UK Ltd
Locations (4):
- United Kingdom (4):
  - Bradford Teaching Hospitals, Bradford
  - Bristol University Hospitals, Bristol
  - Norfolk & Norwich University Hospitals, Norwich
  - University Hospitals Plymouth, Plymouth